CLINICAL TRIAL: NCT00307632
Title: An Open-label Study to Evaluate Contraceptive Efficacy and Safety of the Transdermal Contraceptive System of Norelgestromine and Ethinyl Estradiol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen-Cilag Farmaceutica Ltda. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CR002962; NRGEEPCON4015 (Other: Janssen-Cilag Farmaceutica Ltda.)
Record Dates: First submitted 2006-03-24; First posted 2006-03-28 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2014-05

CONDITIONS: Contraception
Keywords: Contraception; Hormonal patch; Norelgestromine; Ethinyl estradiol

ARMS (1):
- Norelgestromine (NLGM)/Ethinyl Estradiol (EE) (Experimental)
  Interventions: Drug: Norelgestromine (NLGM)/ethinyl estradiol (EE)

INTERVENTIONS:
Drug: Norelgestromine (NLGM)/ethinyl estradiol (EE) — Participants will apply a 20 centimeter square (cm^2) contraceptive transdermal patch on the skin for 1 full week, and then apply a fresh patch for Week 2, and a third patch for Week 3. The fourth week will be patch-free. Each patch delivers 150 microgram (mcg) of NLGM and 20 mcg of EE per day. The treatment duration is of 6 cycles (4 weeks each).

SUMMARY:
The purpose of this study is to evaluate the contraceptive efficacy, safety, cycle control, compliance, and subject satisfaction of the transdermal contraceptive system, norelgestromine and ethinyl estradiol (NLGM / EE).

DETAILED DESCRIPTION:
A multicenter, open label, descriptive study. Five hundred requiring contraception will receive the weekly transdermal contraceptive patch for 6 cycles. At the baseline and after the 1st, 3rd and 6th cycles, satisfaction with the method will be assessed. The contraceptive efficacy will be assessed by the Pearl Index and by life table analysis. To assess satisfaction with the weekly transdermal contraceptive patch, this method will be compared to the previous contraceptive method. Adhesion, cycle control, safety and efficacy are secondary outcomes. Treatment duration: 6 cycles (4 weeks each). The subject will wear a 20 cm2 contraceptive transdermal patch for one full week, apply a fresh patch for week 2, and a third patch for week 3. The fourth week will be patch-free. Each patch deliveries 150 mcg of NLGM and 20 mcg of EE per day.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult females who meet the following selection criteria: Have regular menses occuring every 25-35 days
* Acceptable body mass (< 30) and the weight is < 90 kg
* Has completed her last term pregnancy at least 4 months prior to study admission, is not lactating and has at least one normal menstrual period since her last pregnancy and not breast feeding
* Has a sitting blood pressure systolic < 140 mm/Hg and diastolic < 90 mm/Hg.

Exclusion Criteria:

* Has not received a DepoProvera injection or any other depot hormone injection within six months prior to the screening visit
* Has not used / or in current use of barbiturates, antiepileptics, rifampin, griseofulvin, Hypericum perforatum, or other hepatic enzyme-inducing drugs within 30 days prior to the pre-study visit
* Has not a uncontrolled disorder
* No women over the age 35 who smoke.

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 580 (Actual)
Dates: Start 2003-02; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Pregnancy Rate Determined by Pearl Index | Cycle 6 (Day 168)
  Pearl Index is the number of pregnancies with use of therapy divided by the number of cycles with therapy use. It is an estimation of the number of pregnancies per 100 woman-years of product use.
Pregnancy Rate Determined by Table of Life Analysis | Cycle 6 (Day 168)
  Pregnancy rate was determined by table of life analysis.

SECONDARY OUTCOMES:
Percentage of Participants With Breakthrough Bleeding and/or Spotting | Day 28 of Cycle 1, 3 and 6
  Percentage of participants with breakthrough bleeding and/or spotting was reported.
Compliance Score | Day 28 of Cycle 1, 2, 3, 4, 5 and 6
  Score of compliance was calculated for each participant by dividing the number of cycles with at least one day without the study drug by the total number of therapy cycles. Average score was calculated for cycle 1 to 6.
Percentage of Participants With Response to Satisfaction Questionnaire | Day 28 of Cycle 1, 3 and 6
  Percentage of participants with response to satisfaction questionnaire was reported for following categories: previous contraceptive, method election, physical well-being, emotional well-being, intermenstrual bleeding and intensity, menstrual flow volume, pre-menstrual symptoms, and easiness in ethinyl estradiol and norelgestromin transdermal patch use.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Farmaceutica Ltda. Clinical Trial, Study Director — Janssen-Cilag Farmaceutica Ltda.
Locations (12):
- Brazil (9):
  - Belo Horizonte
  - Botucatu
  - Brasília
  - Curitiba
  - Goiânia
  - Porto Alegre
  - Ribeirão Preto
  - São Paulo
  - Sorocaba
- Mexico (3):
  - Mexico City
  - México
  - Monterrey